CLINICAL TRIAL: NCT04873817
Title: Real-World Outcomes Study on Subjects Treated With Radiofrequency Ablation
Acronym: ROSTRA
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10347
Record Dates: First submitted 2021-05-04; First posted 2021-05-05 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Pain
Keywords: IonicRF™ Generator; ABT-CIP-10347; Radio frequency ablation (RFA); Chronic pain
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- IonicRF Generator and compatible accessories: IonicRF Radiofrequency Generator, along with any country-specific market-released accessory (i.e. electrode, cannula, grounding pad, and adaptor cable) compatible with the IonicRF Generator will be used.
  Interventions: Device: IonicRF Generator and compatible accessories

INTERVENTIONS:
Device: IonicRF Generator and compatible accessories — Participants will receive IonicRF lesion generator, along with any country-specific market-released accessory (i.e. electrode, cannula, grounding pad, and adaptor cable) compatible with the IonicRF Generator

SUMMARY:
ROSTRA is an international, prospective, non-randomized, single-arm, multi-center, and post-market study to collect real-world safety and effectiveness data on Abbott's IonicRF™Generator and compatible RFA accessories. This post-market study is intended to satisfy EU MDR requirements.

ELIGIBILITY:
Inclusion Criteria:

A. All candidate subjects

1. Subject must provide written informed consent prior to any clinical investigation-related procedure
2. Subject is ≥ 18 years of age
3. Subject has chronic pain > 6 months and was unresponsive to conservative management
4. Subject has pain on an NRS scale of ≥ 6
5. Subject is scheduled for an RFA procedure with the IonicRF generator within 30 days of baseline to treat chronic pain at one anatomical region
6. Subject has stable chronic pain medication use for 30 days
7. Subject is willing and able to comply with the prescribed follow-up evaluations

B. Candidate subjects with facet joint pain (lumbar or cervical)

1. Subject has unilateral or bilateral pain on para-spinal palpation and localized pain with extension/lateral bending
2. Subject has facet joint pain confirmed by at least 1 positive medial branch block with 0.5 mL or less of anesthetics (across at least 3 vertebral levels) achieving at least 50% pain relief, with real-time injection of radiographic contrast under fluoroscopic guidance

C. Candidate subjects with sacroiliac joint pain

1. Subject has sacroiliac joint pain based on medical history and physical exam
2. Subject has sacroiliac joint pain confirmed by an infiltration of local anesthetics in the posterior part of the sacroiliac joint achieving at least 50% pain relief

D. Candidate subjects with radicular pain

1. Subject has radicular pain based on medical history and physical exam
2. Subject has radicular pain confirmed by dermatomal mapping corresponding to at least 1 nerve root level

E. Candidate subjects with trigeminal neuralgia

1. Subject has trigeminal pain based on medical history and physical exam
2. Subject did not have any mass effect or stroke causing trigeminal pain confirmed by MRI
3. Subject is ≥ 60 years of age in case of a neurovascular conflict

F. Candidate subjects with knee or hip pain

1. Subject has knee or hip pain based on medical history and physical exam
2. Subject has radiographically confirmed osteoarthritis of the hip or knee, or has chronic pain following joint arthroplasty

Exclusion Criteria:

A. All candidate subjects

1. Subject is currently participating in another clinical investigation that may confound the results of this study.
2. Ongoing systemic or local infection in the area of the procedure.
3. Recent use of anticoagulants or subject with coagulopathy.
4. Primary complaint of deafferentation pain.
5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results.
6. Subject's opioid usage is > 90 morphine equivalents per day.

B. Candidate subjects with trigeminal neuralgia

1. Subject has sensory problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the general chronic pain population referring to the participating pain clinics will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Nura, Edina, Minnesota
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Ainsworth Institute of Pain Management, New York, New York
  - The Spine & Nerve Center of St Francis Hospital, Charleston, West Virginia
- AZ Delta vzw, Roeselare, West Flanders, Belgium
- Hôpital Privé du Confluent, Nantes, Pays de la Loire Region, France
- Germany (2):
  - Krankenhaus Neuwerk Maria von den Aposteln, Mönchengladbach, N. RHIN
  - Universitätsmedizin Berlin - Charité Campus Mitte, Berlin
- Stichting Rijnstate Ziekenhuis - Arnhem, Arnhem, Gelderland, Netherlands
- Spain (2):
  - Hospital Puerta del Mar, Cadiz
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has enrolled 184 subjects at 11 clinical sites in EU and the US. The total duration of the study is expected to be 20 months, including enrollment, data collection from all subjects, and study closeout.
Period: Overall Study
Arm/Group | IonicRF Generator and Compatible Accessories
Started | 184
Completed | 165
Not Completed | 19
Not completed — Subject and/or Family Request Withdrew Consent | 3
Not completed — Lost to Follow-up | 4
Not completed — Unsuccessful RFA Procedure | 1
Not completed — Additional Chronic Pain Treatment for The Same Anatomical Region | 8
Not completed — Other Reasons | 3

BASELINE CHARACTERISTICS:
Population: Subjects who received RF treatment. A total of five enrolled subjects did not receive RF treatment and were considered deregistered.
Arm/Group | IonicRF Generator and Compatible Accessories
Number analyzed (Participants) | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 120
  More than one race | 0
  Unknown or Not Reported | 49
Duration of Chronic Pain (Years) [Mean (Standard Deviation); unit: years] | 9.0 (8.3)
Number of diagnostic blocks provided to participants prior to therapy implementation [Count of Participants; unit: Participants] — A diagnostic block is an injection of a local anesthetic near the area of pain prior to therapy implementation. A favorable response to the diagnostic block (≥50% pain relief) indicates that the nerve is suitable for RF treatment.
  Participants
    1 | 47
    2 | 73
    0 | 59
Pain Relief after the first diagnostic block [Mean (Standard Deviation); unit: units on a scale] — Minimum is 0% and Maximum is 100%.
  units on a scale | 71.9 (18.1)
Pain Relief after second diagnostic block [Mean (Standard Deviation); unit: units on a scale] — Minimum is 0% and Maximum is 100%.
  units on a scale | 74.4 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Relative Change in Numeric Rating Scale (NRS) From Baseline to 3 Months Follow-up Visit
Description: The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their average pain over the past 24 hours specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity. The presented outcome denotes the mean relative change in NRS score, which was defined as (Baseline score - 3-month follow-up visit score)/ Baseline score*100%. Higher scores indicate greater relative pain relief. Minimum value is 0% and maximum value is 100%.
Time Frame: Baseline to 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IonicRF Generator and Compatible Accessories
Number analyzed (Participants) | 162
score on a scale | 34.4 (35.7)
Statistical Analysis 1: Comparison: IonicRF Generator and Compatible Accessories; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Primary Safety Endpoint: Incidence of Device- and Procedure-related Serious Adverse Events
Description: Number of participants with Device- and Procedure-related Serious Adverse Events.
Time Frame: At 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | IonicRF Generator and Compatible Accessories
Number analyzed (Participants) | 162
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 Months
Description: The safety endpoints were evaluated at 3 months follow-up. A total of 162 patients completed 3-month follow-up.
Arm/Group | IonicRF Generator and Compatible Accessories
All-Cause Mortality (participants affected / at risk) | 0/162
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The PI may publish provided that he/she provides the Sponsor with a draft of any Study-related publication, presentation or other disclosure ("Publication") at least sixty (60) calendar days prior to any submission for Sponsor's review
* The PI may not publish the data and results separately from its site until publication of the results of the multi-center study or 18 months after study closure, whichever is sooner.

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT04873817/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT04873817/SAP_001.pdf